CLINICAL TRIAL: NCT02781428
Title: A Multicentre Observational Study Design to Determine the Sensitivity of the UroMark Assay, a Urine Test, to Detect New and Recurrent Low, Intermediate and High Grade Bladder Cancer
Brief Title: To Detect the Sensitivity of the UroMark Assay
Acronym: DETECT II
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0226
Record Dates: First submitted 2016-05-11; First posted 2016-05-24 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective multicentre observational study to assess the sensitivity of the UroMark assay to detect bladder cancer in participants with new or recurrent disease. The study will recruit patients with newly detected or recurrent bladder cancer. The reference standard will be histopathological confirmation of tumour stage and (Ta, T1, ≥T2) and grade 1, 2 or 3 diseases with or without CIS, or CIS alone.

Patients with a visual diagnosis of bladder cancer following cystoscopy will be approached and asked to consent for this study. Consenting participants will be provided with a urine sample collection kit and asked to provide a urine sample. Samples can be provided at home and posted to the receiving lab using the stamped addressed envelope. The urine sample must be obtained before TURBT and following TURBT, patients with NMIBC who require surveillance cystoscopy will be asked to provide a urine sample at 3 monthly intervals for up to 2 years.

The study will be conducted in at least 11 NHS trusts. As DETECT II is an observation study requiring provision of a urine sample, it will be possible for patients in DETECT II to be recruited to other trials.

DETAILED DESCRIPTION:
This study is an observational study and participants will receive the standard of care according to local MDT guidelines for the treatment and surveillance of bladder cancer. As the study involves collection of a urine sample, subjects are permitted to be entered into other trials. The DETECT II study will recruit patients with newly diagnosed and recurrent bladder cancer. As this study is only observational and no intervention is trial related the patients will be given minimum 24 hours to consider this study and decide to take part as they will be approached in clinic at first instance. Due to the initial urine sample being required before any standard of care is received they will be consented within 24 hours of being informed of the study. Most newly diagnosed bladder cancers are detected in patients being investigated for haematuria and attending a haematuria clinic. Most recurrent bladder cancers are detected by cystoscopy at bladder cancer check cystoscopy clinics.

Patients with a visual diagnosis or new or recurrent bladder cancer will be eligible for the DETECT II study. The baseline UroMark urine collection will be collected once the visual diagnosis of bladder cancer is established. The UroMark sample must be provided before TURBT in all cases.

Patients will be approached following cystoscopy and asked to consent to study entry. The DETECT II study will involve obtaining a voided urine sample. Patients will be given a UroMark urine sample kit and asked to provide the urine sample at home and post the sample to the receiving lab using the stamped addressed envelope.

Patients will receive the standard tests and investigations for bladder cancer. The standard treatment for bladder cancer is summarised as:

* TURBT following which it is recommended that patients with NMIBC receive a single instillation of chemotherapy unless contraindicated.
* Intermediate risk NMIBC will be considered for a 6 week inductive course of intravesical chemotherapy after TURBT.
* High risk NMIBC may require a second TURBT called re-resection TURBT, usually within 6 weeks of the first. The re--resection or second TURBT is performed for pathological stage pT1 tumours to exclude residual detrusor muscle invasion (stage pT2 at least). There are 2 treatment choices when the high risk status has been confirmed clinically:
* A course of inductive followed by maintenance intravesical BCG
* An operation to remove the bladder (a cystectomy).
* Cystectomy or radiotherapy are the options for patients diagnosed with MIBC

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 years of age.
* Visual diagnosis or suspected diagnosis of bladder cancer following cystoscopy.
* Able to give informed written consent to participate

Exclusion Criteria:

* Unwilling to undergo TURBT
* Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DETECT II will recruit patients attending haematuria clinics, check cystoscopy clinics or at pre-assessment clinic prior to TURBT. All patients who have a visual diagnosis of new or recurrent bladder cancer after flexible cystoscopy can be approached.
Sampling Method: Non-Probability Sample
Enrollment: 1643 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
The sensitivity of the UroMark assay to detect bladder cancer for grades 1-3, stage Ta -T4 | 2 years

SECONDARY OUTCOMES:
The ability of the UroMark assay to detect the recurrence in NMIBC in patients undergoing cystoscopic surveillance for bladder cancer | 2 years
A comparison between UroMark and other control assays including molecular tests | 2 years

CONTACTS AND LOCATIONS:
Locations (19):
- United Kingdom (19):
  - Tameside General Hospital, Ashton-under-Lyne
  - East Lancashire Hospitals NHS Trust, Blackburn
  - Royal Bolton Hospital, Bolton
  - The Pennine Acute Hospitals NHS Trust, Bury
  - University Hospital Coventry, Coventry
  - Medway Maritime Hospital, Gillingham
  - University College London Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - Macclesfield Hospital, Macclesfield
  - Norfolk & Norwich University Hospital, Norwich
  - King's Mill Hospital, Nottingham
  - East Surrey Hospital, Redhill
  - Northern Lincolnshire & Goole NHS Foundation Trust, Scunthorpe
  - Western Sussex Hospitals NHS Foundation Trust, Shoreham-by-Sea
  - Royal Shrewsbury Hospital, Shrewsbury
  - Stepping Hill Hospital, Stockport
  - University Hospital of North Tees, Stockton-on-Tees
  - Royal Albert Edward Infirmary, Wigan
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Papers will be prepared for publication in general and urological peer-reviewed journals. The findings will also be presented at national and international conferences. The results of the study will be disseminated regardless of the direction of effect. Authorship will be determined according to an agreed Publication Policy.

REFERENCES:
- [Derived] Tan WS, Teo CH, Chan D, Ang KM, Heinrich M, Feber A, Sarpong R, Williams N, Brew-Graves C, Ng CJ, Kelly J; DETECT II trial collaborators. Exploring patients' experience and perception of being diagnosed with bladder cancer: a mixed-methods approach. BJU Int. 2020 May;125(5):669-678. doi: 10.1111/bju.15008. Epub 2020 Feb 12. PMID 31975539
- [Derived] Tan WS, Teo CH, Chan D, Heinrich M, Feber A, Sarpong R, Allan J, Williams N, Brew-Graves C, Ng CJ, Kelly JD; DETECT II trial collaborators. Mixed-methods approach to exploring patients' perspectives on the acceptability of a urinary biomarker test in replacing cystoscopy for bladder cancer surveillance. BJU Int. 2019 Sep;124(3):408-417. doi: 10.1111/bju.14690. Epub 2019 Mar 4. PMID 30694612
- [Derived] Tan WS, Feber A, Dong L, Sarpong R, Rezaee S, Rodney S, Khetrapal P, de Winter P, Ocampo F, Jalil R, Williams NR, Brew-Graves C, Kelly JD. DETECT I & DETECT II: a study protocol for a prospective multicentre observational study to validate the UroMark assay for the detection of bladder cancer from urinary cells. BMC Cancer. 2017 Nov 15;17(1):767. doi: 10.1186/s12885-017-3758-7. PMID 29141603